CLINICAL TRIAL: NCT02991469
Title: An Open-label, Sequential, Ascending, Repeated Dose-finding Study of Sarilumab, Administered With Subcutaneous (SC) Injection, in Children and Adolescents, Aged 1 to 17 Years, With Systemic Juvenile Idiopathic Arthritis (sJIA), Followed by an Extension Phase
Brief Title: A Repeated Dose-finding Study of Sarilumab in Children and Adolescents With Systemic Juvenile Idiopathic Arthritis (SKYPS)
Acronym: SKYPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRI13926; U1111-1177-3584 (Registry Identifier: ICTRP); 2024-512701-11 (Registry Identifier: CTIS)
Record Dates: First submitted 2016-10-14; First posted 2016-12-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sarilumab (Experimental): Participants will receive one of two ascending doses (or an additional intermediate dose based on available data) of sarilumab by subcutaneous (SC) injection based on body weight. All the participants will receive the selected dose once the selected dose is identified. Sarilumab will be given during 12-week core treatment phase followed by a 144- week extension treatment phase.
  Interventions: Drug: Sarilumab SAR153191 (REGN88)

INTERVENTIONS:
Drug: Sarilumab SAR153191 (REGN88) — Pharmaceutical form: Solution
  Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To describe the pharmacokinetic (PK) profile of sarilumab in patients aged 1-17 years with Systemic Juvenile Idiopathic Arthritis (sJIA) in order to identify the dose and regimen for adequate treatment of this population.

Secondary Objective:

To describe the pharmacodynamics (PD) profile, the efficacy, and the long term safety of sarilumab in patients with sJIA.

DETAILED DESCRIPTION:
The total study duration per patient will be 166 weeks that will consist of a 4- week screening, a 12-week core treatment phase, a 144-week extension phase, and a 6-week post-treatment follow-up.

ELIGIBILITY:
Inclusion criteria :

* Male and female patients aged ≥1 and ≤17 years (or country specified age requirement, ≥6 to ≤17 years for Russia) at the time of the screening visit.
* Diagnosis of systemic JIA subtype according to the International Associations against Rheumatism (ILAR) 2001 Juvenile Idiopathic Arthritis (JIA) Classification Criteria OR According to 2024 EULAR/PReS recommendation at Screening.
* Patient with an inadequate response to current treatment and considered as a candidate for a biologic disease modifying anti rheumatic drug (DMARD) as per investigator's judgment.

Exclusion criteria:

* Body weight <10 kg or >60 kg for patients enrolled in the ascending dose cohorts, then body weight <10 kg for patients subsequently enrolled at the selected dose.
* Uncontrolled severe systemic symptoms and/or Macrophage Activation Syndrome (MAS) within 6 months prior to screening.
* History of or ongoing interstitial lung disease, pulmonary hypertension, pulmonary alveolar proteinosis.
* If nonsteroidal anti-inflammatory drugs (NSAIDs) (including cyclo oxygenase-2 inhibitors [COX-2]) taken, dose stable for less than 2 weeks prior to the baseline visit and/or dosing prescribed outside of approved label.
* If non-biologic DMARD taken, dose stable for less than 6 weeks prior to the baseline visit or at a dose exceeding the recommended dose as per local labeling.
* If oral glucocorticoid taken, dose exceeding equivalent prednisone dose 1 mg/kg/day (or 60 mg/day) within 3 days prior to baseline.
* Use of parenteral or intra-articular glucocorticoid injection within 4 weeks prior to baseline.
* Prior treatment with anti-interleukin 6 (IL-6) or IL-6 receptor (IL-6R) antagonist therapies, including but not limited to tocilizumab or sarilumab.
* Treatment with any biologic treatment for sJIA within 5 half-lives prior to the first dose of sarilumab (the required off treatment periods and procedures may vary according to local requirements).
* Treatment with a Janus kinase inhibitor within 4 weeks prior to the first dose of sarilumab; and treatment with growth hormone within 4 weeks prior to the first dose of sarilumab (the required off treatment periods and procedures may vary according to local requirements).
* Treatment with any investigational biologic or non-biologic product within 8 weeks or 5 half-lives prior to baseline, whichever is longer.
* Exclusion related to tuberculosis.
* Exclusion criteria related to past or current infection other than tuberculosis.
* Any live, attenuated vaccine within 4 weeks prior to the baseline visit, such as varicella-zoster, oral polio, rubella vaccines. Killed or inactive vaccine may be permitted based on the Investigator's judgment.
* Exclusion related to history of a systemic hypersensitivity reaction to any biologic drug and known hypersensitivity to any constituent of the product.
* Laboratory abnormalities at the screening visit (identified by the central laboratory).
* Severe cardiac disease due to sJIA.
* Pregnant or breast-feeding female adolescent patients.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
Assessment of PK parameter: maximum serum concentration observed (Cmax) | Up to Week 12
Assessment of PK parameter: Area under the serum concentration versus time curve calculated using the trapezoidal method during a dose interval (AUC0-t) | Up to Week 12
Assessment of PK parameter: Concentration observed before treatment administration during repeated dosing (Ctrough) | Up to Week 12

SECONDARY OUTCOMES:
Number of patients with adverse events | Core treatment phase: Up to Week 12. Extension phase: Up to Week 162
Proportion of participants with local reactions after injection | Core treatment phase: Up to Week 12. Extension phase: Up to Week 156
Proportion of participants with Investigator Global Assessment (IGA) of disease activity below a defined value on 1-100 VAS scale | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
Proportion of participants with Parent / patient Global Assessment (PGA) of well-being below a defined value on 1-100 VAS scale | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
Proportion of participants with clinically inactive disease (CID) | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
Changes in glucocorticoid use | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
Juvenile Idiopathic Arthritis ACR30/50/70/90/100 (in the absence of fever) response rate | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
  Population according to the 2001 ILAR classification
Change from baseline in individual JIA ACR components | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
  Population according to the 2001 ILAR classification
Change from baseline in Systemic Juvenile Arthritis Disease Activity Score-10 (sJADAS-10) | Core treatment phase: Up to Week 12. Extension phase: At weeks 24, 48, and every 24 weeks up to Week 156
  Population according to the 2001 ILAR classification
Assessment of participants with disease-related symptoms | At Week 4
  Population according to the 2024 EULAR / PReS
Changes in IL-6 associated biomarkers | Up to Week 12
  Population according to the 2001 ILAR classification and the 2024 EULAR / PReS

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (28):
- Investigational Site Number : 0320004, San Miguel de Tucumán, Tucumán Province, Argentina
- Investigational Site Number : 1240110, Calgary, Alberta, Canada
- Investigational Site Number : 2460040, Helsinki, Finland
- France (3):
  - Investigational Site Number : 2500041, Bron
  - Investigational Site Number : 2500042, Montpellier
  - Investigational Site Number : 2500040, Paris
- Germany (5):
  - Investigational Site Number : 2760064, Berlin
  - Investigational Site Number : 2760065, Berlin
  - Investigational Site Number : 2760062, Hamburg
  - Investigational Site Number : 2760060, Sankt Augustin
  - Investigational Site Number : 2760063, Sendenhorst
- Investigational Site Number : 3720001, Crumlin, Dublin, Ireland
- Italy (3):
  - Investigational Site Number : 3800051, Genoa, Genova
  - Investigational Site Number : 3800054, Milan, Milano
  - Investigational Site Number : 3800052, Rome, Roma
- Russia (4):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430062, Moscow
  - Investigational Site Number : 6430063, Moscow
  - Investigational Site Number : 6430065, Ufa
- Spain (6):
  - Investigational Site Number : 7240055, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240050, Esplugues de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240053, Madrid
  - Investigational Site Number : 7240056, Madrid
  - Investigational Site Number : 7240054, Málaga
  - Investigational Site Number : 7240051, Valencia
- United Kingdom (3):
  - Investigational Site Number : 8260031, London, London, City of
  - Investigational Site Number : 8260034, Leeds
  - Investigational Site Number : 8260033, Liverpool

REFERENCES:
- See also: DRI13926 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26032&tenant=MT_SNY_9011